CLINICAL TRIAL: NCT01726686
Title: Evaluation of Intra-articular Continuous Infusion Pump With Ropivacaine in Addition to Local Infiltration Analgesia (LIA) in Total Knee Arthroplasty (TKA). A Placebo Controlled Randomised Trial.
Brief Title: Pain Treatment After TKA With LIA and Intra-articular Continuous Infusion Pump
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Principal Investigator, Gunnar Flivik, Associate Professor, MD PhD, Region Skane
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LIA-Pump_AA
Record Dates: First submitted 2012-10-30; First posted 2012-11-15 (Estimated); Last update posted 2014-11-26 (Estimated); Status verified 2014-11

CONDITIONS: Postoperative Pain Management
Keywords: Total Knee Arthroplasty
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ropivacaine in the pump (Active Comparator): The intra-articular Continuous Infusion Pump is filled with Ropivacaine,10 mg/ml, set at 2 ml/hour for 48 hours postoperatively.
  Interventions: Drug: Ropivacaine
- Placebo in the pump (Placebo Comparator): The intra-articular Continuous Infusion Pump is filled with NaCl, set at 2 ml/hour for 48 hours postoperatively.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ropivacaine — 100 ml Ropivacaine 10mg/ml in a continuous infusion pump set at 2 ml/hour
  Other Names: Naropin, Narop
  Arms: Ropivacaine in the pump
Drug: Placebo
  Arms: Placebo in the pump

SUMMARY:
The purpose of this study is to evaluate the effect on postoperative pain and function by adding intraarticular continuous infusion pump with local anesthetic after total knee arthroplasty where local infiltration analgesia has already been given.

DETAILED DESCRIPTION:
200 patients with osteoarthritis (OA) of the knee necessitating total knee arthroplasty are entered into the study. All patients are given a standard protocol of analgesics pre- and postoperatively. All patients get periarticular LIA-injection (150 ml) with a total of 300 mg Ropivacaine, 30 mg Toradol and 0.5 mg Adrenalin. In the end of the operation all patients get an epidural type of catheter intraarticular with a coupled continuous infusion pump that delivers 2 ml per hour and are disconnected after 48 hours. The University hospital pharmacy has prepared 200 pumps; 100 Active substance pumps with 100 ml Ropivacaine (10mg/ml) and 100 placebo pumps with 100 ml sodium chloride (NaCl). All patients are by computer software randomized to receive either active or placebo pump. Only one nurse, not involved in neither the operation nor the after treatment, has the key to what substance it is in the numbered pumps. Thus, it is a double blinded trial during the whole follow up period. Before the operation the patients are asked to fill out a knee specific outcome questionnaire, the Knee injury and Osteoarthritis Outcome Score (KOOS), and a general outcome questionnaire, the Euroqol (EQ-5D), and the knee range of motion is measured by a physiotherapist. After the operation the patients are monitored at the ward by the nurses and physiotherapists. The level of pain is measured twice daily (noon and 8 PM) according to the Visual-Analog-Scale (VAS). The range of motion and is measured on day 4 and at the day 14 and day 30 follow up. The number of days the patients need to stay in hospital after operation are registered. The amount of extra doses of analgesics the patient requires are registered as well as the complications (illness, wound problems, infections etc). The patients are to be followed clinically for 2 years as well as with outcome questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Primary osteoarthritis of the knee necessitating total knee replacement
* Patients who understand the conditions of the study and are willing to participate for the length of the prescribed follow-up

Exclusion Criteria:

* Known allergy to local anaesthetics or other contraindication for the use of local anaesthetics.
* Treatment with Warfarin.
* Bilateral operation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2010-02; Primary Completion 2011-07 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Change in postoperative pain | The first 4 postoperative days at noon and 8 PM
  The patient are asked to grade their pain on a VAS-scale (0-100)twice daily for the first 4 days after the TKA operation and at the 2 weeks follow-up. Changes in pain during this time frame are recorded to see if there are any differences between the two groups.

SECONDARY OUTCOMES:
Extra oral analgesia consumption | First 4 postoperative days
  All extra analgesia consumption are noted during the first 4 postoperative days. All patients have a standard pain management medication (depending on weight, age and sex) and only extra doses are noted.

OTHER OUTCOMES:
Number of postoperative days in hospital | Duration of hospital stay, an expected time frame of 4-5 days
  The number of days the patient needs to stay in hospital after operation are noted
Pre- and postoperative knee range of motion | At preoperative admission for operation (about 2 weeks prior), day 4, 14 and 30 postoperatively
  The range of motion in the affected knee are registered with a goniometer at the preoperative admission for operation, about 2 weeks prior to the operation and then on day 4, 14 and 30 postoperatively.
Postoperative complications | 2 years postoperatively
  All complications postoperatively are registered for the first 2 years.
Knee specific and general questionaire | preoperatively (about 2 weeks prior to op), 1 and 2 years postoperatively
  The patients are asked to fill out the general health questionaire EQ-5D as well as the knee specific questionaire KOOS preoperatively at the admission for surgery (about 2 weeks before the operation) and at 1 and 2 year follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar Flivik, MD PhD, Principal Investigator — Dept of Orthopedics, Skane University Hospital, Lund University, Sweden
Locations (1):
- Department of Orthopedics, Skane University Hospital, Lund University, Lund, Sweden